CLINICAL TRIAL: NCT07354321
Title: Thrombo-inflammation Des Maladies Neurovascualires aiguës : définition de Nouvelles Cibles thérapeutiques (TARGETS)
Brief Title: Thrombo-inflammation in Acute Neurovascular Diseases: Definition of New Therapeutic Targets (TARGETS)
Status: Not yet recruiting | Type: Observational
Sponsor: François Delvoye (Other)
Responsible Party: Sponsor-Investigator, François Delvoye, Doctor, Centre Hospitalier Universitaire de Liege
Organization: Centre Hospitalier Universitaire de Liege (Other)
Other Study IDs: B7072025000062
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Delayed Cerebral Ischemia After Subarachnoid Hemorrhage; Ischemic Stroke of Large or Medium Vessels
Keywords: delayed cerebral ischemia; subarachnoid hemorrhage; ischemic stroke
MeSH Terms: conditions — Subarachnoid Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AIC: Patient with rapid progression of necrotic volume after an ischemic stroke due to large- or medium-vessel occlusion in the anterior circulation
- HSA: Patient with delayed cerebral ischemia after subarachnoid hemorrhage
- healthy volunteer: healthy volunteer

SUMMARY:
The objective of this observational study is to compare the relative concentrations of various thrombo-inflammatory markers at different follow-up time points in:

* patients with or without delayed cerebral ischemia after subarachnoid hemorrhage, and
* patients with or without rapid progression of necrotic volume after an ischemic stroke due to large- or medium-vessel occlusion in the anterior circulation.

The main question this study aims to answer is: How do thrombo-inflammatory marker concentrations evolve over time and differ between patients? Researchers will compare patients with or without delayed cerebral ischemia after subarachnoid hemorrhage, as well as patients with or without rapid progression of necrotic volume following an ischemic stroke due to large- or medium-vessel occlusion in the anterior circulation, to determine whether there are differences in thrombo-inflammatory marker concentrations and in their evolution over time.

Participants will undergo blood sampling at five different time points. In addition, participants will complete a Montreal Cognitive Assessment (MoCA) questionnaire during the 3-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Admitted within 8 hours of an acute ischemic stroke (AIS) due to large-vessel occlusion (LVO) or medium-vessel occlusion (MeVO) of the anterior circulation, with a NIHSS (National Institutes of Health Stroke Scale) score > 5 (M1, M2, M3, A1, A2, A3, P1, P2)
* Or admitted within 36 hours of acute symptoms related to aneurysmal subarachnoid hemorrhage (SAH)

Exclusion Criteria:

* Patients with pre-existing functional and/or cognitive disability (modified Rankin Scale, mRS > 1)
* Patients under legal protection or guardianship
* Patients with secondary hemorrhagic transformation of an acute ischemic stroke

Patients with acute ischemic stroke and NIHSS > 5 without LVO or MeVO of the anterior circulation on imaging will be secondarily excluded. Perfusion imaging will not be performed as part of the research protocol. Excluded patients will be replaced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Among patients treated at Liège University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2032-05 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Investigation of changes in thrombo-inflammatory marker concentrations between patients and over time. | From enrollment to Month 3 visit
  Investigation of changes in thrombo-inflammatory marker concentrations between patients and over time.

IPD SHARING:
Plan to Share IPD: Undecided
Accessible upon request after publication

REFERENCES:
- [Background] Gatti JL, Dacheux JL. Immunological cross-reaction between sperm dynein heavy chains from different species. Reprod Nutr Dev. 1996;36(2):213-20. doi: 10.1051/rnd:19960206. PMID 8663918
- [Background] Lewis DF. Quantitative structure-activity relationships in a series of alcohols exhibiting inhibition of cytochrome P-450-mediated aniline hydroxylation. Chem Biol Interact. 1987;62(3):271-80. doi: 10.1016/0009-2797(87)90027-5. PMID 3621372
- [Background] Rector TS, Carlyle PF, Cohn JN. Reduced atrial natriuretic factor after ligation of the left coronary artery in rats. Am Heart J. 1985 Dec;110(6):1197-9. doi: 10.1016/0002-8703(85)90012-2. PMID 2933941
- [Background] Knaff DB. Structure and regulation of ribulose-1,5-bisphosphate carboxylase/oxygenase. Trends Biochem Sci. 1989 May;14(5):159-60. doi: 10.1016/0968-0004(89)90264-8. No abstract available. PMID 2773037
- [Background] Liu X, Wang CA, Chen YZ. [Bovine serum albumin-conjugated corticosterone inhibits the release of arginine vasopressin]. Sheng Li Xue Bao. 1996 Apr;48(2):173-8. Chinese. PMID 9389169
- [Background] Hayes JC. Practice improvement project measures radiology quality. Diagn Imaging (San Franc). 1999 Feb;21(2):22. No abstract available. PMID 10351546
- [Background] Fujisawa T, Ikegami H, Yamato E, Takekawa K, Nakagawa Y, Hamada Y, Oga T, Ueda H, Shintani M, Fukuda M, Ogihara T. Association of Trp64Arg mutation of the beta3-adrenergic-receptor with NIDDM and body weight gain. Diabetologia. 1996 Mar;39(3):349-52. doi: 10.1007/BF00418352. PMID 8721782
- [Background] Angra SK, Mohan M, Saini JS. Medical therapy of cataract (evaluation of Catalin). Indian J Ophthalmol. 1983 Jan;31(1):5-8. No abstract available. PMID 6354928
- [Background] Boll IT, Domeyer C. Lymphocytes as inducers of mitoses of human morphologically identifiable progenitor cells. Phase contrast observations. Exp Hematol. 1982 Apr;10(4):326-31. PMID 7047181
- [Background] Coulibaly AP, Pezuk P, Varghese P, Gartman W, Triebwasser D, Kulas JA, Liu L, Syed M, Tvrdik P, Ferris H, Provencio JJ. Neutrophil Enzyme Myeloperoxidase Modulates Neuronal Response in a Model of Subarachnoid Hemorrhage by Venous Injury. Stroke. 2021 Oct;52(10):3374-3384. doi: 10.1161/STROKEAHA.120.033513. Epub 2021 Aug 18. PMID 34404234
- [Background] Ishikawa M, Kajimura M, Morikawa T, Tsukada K, Tsuji T, Kusaka G, Tanaka Y, Suematsu M. Leukocyte plugging and cortical capillary flow after subarachnoid hemorrhage. Acta Neurochir (Wien). 2016 Jun;158(6):1057-67. doi: 10.1007/s00701-016-2792-6. Epub 2016 Apr 4. PMID 27040552
- [Background] Ishikawa M, Kusaka G, Yamaguchi N, Sekizuka E, Nakadate H, Minamitani H, Shinoda S, Watanabe E. Platelet and leukocyte adhesion in the microvasculature at the cerebral surface immediately after subarachnoid hemorrhage. Neurosurgery. 2009 Mar;64(3):546-53; discussion 553-4. doi: 10.1227/01.NEU.0000337579.05110.F4. PMID 19240618
- [Background] Sehba FA, Mostafa G, Friedrich V Jr, Bederson JB. Acute microvascular platelet aggregation after subarachnoid hemorrhage. J Neurosurg. 2005 Jun;102(6):1094-100. doi: 10.3171/jns.2005.102.6.1094. PMID 16028769
- [Background] Chen Y, Galea I, Macdonald RL, Wong GKC, Zhang JH. Rethinking the initial changes in subarachnoid haemorrhage: Focusing on real-time metabolism during early brain injury. EBioMedicine. 2022 Sep;83:104223. doi: 10.1016/j.ebiom.2022.104223. Epub 2022 Aug 13. PMID 35973388
- [Background] Hoh BL, Ko NU, Amin-Hanjani S, Chou SH-Y, Cruz-Flores S, Dangayach NS, Derdeyn CP, Du R, Hanggi D, Hetts SW, Ifejika NL, Johnson R, Keigher KM, Leslie-Mazwi TM, Lucke-Wold B, Rabinstein AA, Robicsek SA, Stapleton CJ, Suarez JI, Tjoumakaris SI, Welch BG. 2023 Guideline for the Management of Patients With Aneurysmal Subarachnoid Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2023 Jul;54(7):e314-e370. doi: 10.1161/STR.0000000000000436. Epub 2023 May 22. PMID 37212182